CLINICAL TRIAL: NCT03936634
Title: An Innovative Approach Towards Understanding and Arresting Type 1 Diabetes (INNODIA)
Acronym: INNODIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cambridge (Other)
Collaborators: Innovative Medicines Initiative (Other); Juvenile Diabetes Research Foundation (Other); The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Principal Investigator, David Dunger, Professor of Paediatrics, University of Cambridge
Other Study IDs: INNODIA 01; 210497 (Other: IRAS Project ID); 115797 (Other Grant/Funding Number: Innovative Medicines Initiative)
Record Dates: First submitted 2019-03-21; First posted 2019-05-03 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Observation study; First degree relatives; Beta cell; C-Peptide; Immune cells; Disease progression
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Serum, plasma, whole blood, urine, stool, dried blood spot
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Newly Diagnosed (ND): Recruited within 6 weeks of type 1 diabetes diagnosis. Age between 1 and <45 years
- Unaffected Family members (UFM): Participants who are not diabetic but have a first degree relative with type 1 diabetes diagnosed < 45 years of age.
  Age between 1 and <45 years

SUMMARY:
INNODIA is a global consortium linking 26 academic institutions, 4 industrial partners, a small to medium enterprise (SME), and 2 patient organisations, bringing their knowledge and experience together with one common goal: "To fight type 1 diabetes". (www.innodia.eu).

The project, approved in November 2015 and launched in January 2016, runs under the framework of the Innovative Medicines Initiative - Joint Undertaking (https://www.imi.europa.eu/projects-results/project-factsheets/innodia) with a dedicated governance structure ensuring close interaction, communication and adherence to the objectives and deliverables of the consortium.

The overall aim of INNODIA is to advance in a decisive way how to predict, stage, evaluate and prevent the onset and progression of type 1 diabetes (T1D). For this, INNODIA has established a comprehensive and interdisciplinary network of clinical and basic scientists, who are leading experts in the field of T1D research in Europe, with complementary expertise from the areas of immunology, Beta-cell biology, biomarker research and T1D therapy, joining forces in a coordinated fashion with industry partners and two foundations, as well as with all major stakeholders in the process, including regulatory bodies and patients with T1D and their families.

One of the objectives of INNODIA is to develop a new European clinical research network with standardized protocol based on repeated measures of C-peptide (including home measurements) and comprehensive collection of appropriate biological samples for 'omics', immune, viral and microbiome studies in new onset T1D patients and high-risk auto-antibody positive subjects. A protocol for the harmonization of sample collections in newly diagnosed type 1 diabetic patients and first degree relatives of patients with type 1 diabetes was developed following extensive preliminary work involving partners from across all specialities. Core laboratories with experience in their respective field were set up for analysis of auto-antibodies, fresh immune cells, handling of frozen immune cells, C-peptide measures. A series of standard operating procedures for sample collections and analysis were agreed. Sample tracking between clinical centres and central laboratories was included into a purposely designed electronic case report form (eCRF) into which all clinical and laboratory data collected are captured.

DETAILED DESCRIPTION:
This is a longitudinal observational study of the relationship between measures of β-cell function, genotype, immunological phenotype and potential environmental factors over time, in individuals with new onset T1D or first degree relatives at higher risk for T1D due to the presence of auto-antibodies.

It is a multicentre international study involving clinical centres across Europe which is unique in the following ways:

1. The first such collaboration in Europe
2. Novel evaluation of C-peptide/β-cell function using both home dried blood spots and regular hospital mixed meal tolerance tests or oral glucose tolerance tests
3. Identical study procedures across all clinical centres
4. Centralised analysis/storage of clinically relevant samples
5. The creation of a living 'Biobank' whereby participants can be recalled for study on the basis of specific genotype/phenotypes
6. Linkage to innovative study of novel biomarkers to inform future interventional strategies
7. A potential pipeline for future recruitment and consent to novel innovative interventional strategies

The study is divided into 2 arms:

In arm A, the investigators plan to recruit 1500 newly diagnosed T1D patients within 6 weeks from diagnosis. The last study visit will be planned 2 years from diagnosis or until the end of the study. Therefore, the duration of the study will be approximately 2 years consisting of 5 visits. At baseline, C-peptide and immunophenotyping are evaluated. Follow up consists of regular mixed meal tolerance test (MMTT) and providing blood, urine and stool samples for 'omics', immune, viral and microbiome studies. Home dried blood spots (DBS) pre and post a standardized meal will be collected monthly for the duration of the study.

These recruited participants will be included for further observational study, confirmation of potential biomarkers and will ultimately provide a pipeline for future recruitment to interventional studies.

In arm B, the investigators plan to screen approximately 4500 unaffected first degree family members across all centres during the first 3 years. The family members will be screened for 4 auto-antibodies (GAD65, IA-2A, IAA, ZnT8A).

Unaffected family members who are auto-antibody positive will be followed up for approximately 4 years consisting of visits every 6 months for the first 2 years and then every 12 months until the end of the study. Follow up will consist of regular oral glucose tolerance test (OGTT) and providing blood, urine and stool samples for 'omics', immune, viral and microbiome studies. Home dried blood spots (DBS) will be collected monthly for the duration of the study.

Unaffected participants who are auto-antibody negative will be sent annual questionnaires until the end of the study.

All study participants will be consented to a living 'Biobank' where we will be able to request participants to be recalled by genotype/phenotype for further studies involving blood, urine and stool samples.

ELIGIBILITY:
Newly diagnosed:

Inclusion Criteria:

* Have given written informed consent to participate.
* Be aged between 1 year and <45 years.
* Less than 6 weeks from diagnosis of type 1 diabetes and requiring insulin treatment.

Exclusion Criteria:

* Non-type 1 diabetes (type 2, monogenic diabetes and secondary diabetes)
* Concurrent use of long term immunosuppressive agents including oral steroids or medication likely to confound the interpretation of study results.
* Expected non-compliance with the protocol.
* Any medical history or clinical relevant abnormality that is deemed by the principal investigator and/or co-investigator to make the patient ineligible for inclusion because problems in interpreting data or safety concern.
* Participating in interventional or other drug research studies which could affect the primary objectives of the study.

Unaffected Family Members:

Inclusion Criteria:

* Have given written informed consent to participate.
* Be aged between 1 year and <45 years.
* Have a first degree relative with type 1 diabetes (parent, child, full or half siblings) diagnosed <45 years of age

Exclusion Criteria:

* The affected first degree relative has type 2 diabetes, monogenic diabetes or diabetes secondary to another medical condition.
* Concurrent use of long term immunosuppressive agents including oral steroids or medication likely to confound the interpretation of study results.
* Expected non-compliance with the protocol.
* Any medical history or clinical relevant abnormality that is deemed by the principal investigator and/or co-investigator to make the patient ineligible for inclusion because problems in interpreting data or safety concern.
* Participating in interventional or other drug research studies which could affect the primary objectives of the study.

Ages: 1 Year to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Newly diagnosed patients with Type 1 diabetes.
  Unaffected first degree family members of patients with type 1 diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2016-11-14 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Arm A - Newly Diagnosed people with Type 1 diabetes | 24 months
  Rate of decline in Beta cell function as assessed by mixed meal tolerance test and home dried blood spot C-peptide measures over the first 24 months from diagnosis of Type 1 diabetes.
Arm B - Auto-antibody positive first degree family members | 48 months
  Development of diabetes as defined by the American Diabetes Association in auto-antibody positive family members followed longitudinally.

SECONDARY OUTCOMES:
Arm A - Newly diagnosed patients with Type 1 diabetes | 24 months
  Changes in HbA1c, insulin dose, autoantibody levels over the first 24 months from diagnosis.
Arm A - Newly diagnosed patients with Type 1 diabetes - Systematic evaluation of biological samples | 24 months
  Systematic evaluation of biological samples using multiple 'omics' approach to identify biomarkers which predict rate of deterioration in C-peptide measures
Arm A - Newly diagnosed patients with Type 1 diabetes - Framework | 24 months
  To develop a robust observational framework for future interventional studies.
Arm B - Auto-antibody positive first degree family members - glucose tolerance | 48 months
  Changes in glucose tolerance as determined by repeated oral glucose tolerance tests over the follow up period of 48 months
Arm B - Auto-antibody positive first degree family members - Systematic evaluation of biological samples | 48 months
  Systematic evaluation of biological samples, using multiple 'omics' approach, auto antibodies to identify biomarkers which predict rate of progression to diabetes.
Arm B - Auto-antibody positive first degree family members - Framework | 48 months
  Developing a robust framework for future interventional studies.

CONTACTS AND LOCATIONS:
Overall Officials: David B Dunger, Principal Investigator — University of Cambridge; Mikael Knip, Principal Investigator — University of Helsinki; Chantal Mathieu, Study Chair — Katholieke Universteit Leuven
Locations (19):
- Medical University of Graz, Graz, Austria
- Belgium (2):
  - Universitee Libre de Bruxelles, Brussels
  - Katholieke Universiteit Leuven, Leuven
- University of Copenhagen, Copenhagen, Denmark
- Finland (3):
  - University of Helsinki, Helsinki
  - University of Oulu, Oulu
  - Turku University Hospital, Turku
- Institut National de la Sante et de la Recherche Medicale (INSERM), Paris, France
- Germany (2):
  - Children's Hospital Auf der Bult, Hannover Medical School, Hanover
  - University of Ulm, Ulm
- Italy (3):
  - San Raffaele Hospital, Milan
  - Ospedale Pediatrico Bambino Gesu, Rome
  - University of Studi di Siena, Siena
- University of Luxembourg, Luxembourg, Luxembourg
- Oslo Universitetssytehus HF, Oslo, Norway
- Medical University of Silesia Katowice, Katowice, Poland
- University of Ljubljana, Ljubljana, Slovenia
- University of Lund, Malmo, Sweden
- University of Cambridge, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andellini M, Haleem S, Angelini M, Ritrovato M, Schiaffini R, Iadanza E, Pecchia L. Artificial intelligence for non-invasive glycaemic-events detection via ECG in a paediatric population: study protocol. Health Technol (Berl). 2023;13(1):145-154. doi: 10.1007/s12553-022-00719-x. Epub 2023 Jan 23. PMID 36761922
- [Derived] Wilhelm-Benartzi CS, Miller SE, Bruggraber S, Picton D, Wilson M, Gatley K, Chhabra A, Marcovecchio ML, Hendriks AEJ, Morobe H, Chmura PJ, Bond S, Aschemeier-Fuchs B, Knip M, Tree T, Overbergh L, Pall J, Arnaud O, Haller MJ, Nitsche A, Schulte AM, Mathieu C, Mander A, Dunger D. Study protocol: Minimum effective low dose: anti-human thymocyte globulin (MELD-ATG): phase II, dose ranging, efficacy study of antithymocyte globulin (ATG) within 6 weeks of diagnosis of type 1 diabetes. BMJ Open. 2021 Dec 7;11(12):e053669. doi: 10.1136/bmjopen-2021-053669. PMID 34876434